CLINICAL TRIAL: NCT00549731
Title: Database for Persons Interested in Research Studies of Developmental Disorders
Brief Title: Participant Database for Autism Research Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Tal Kenet, Associate Professor, Massachusetts General Hospital
Other Study IDs: 2007-P-000062; 5R01MH117998 (NIH)
Record Dates: First submitted 2007-10-15; First posted 2007-10-26 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; autistic; language; development; developmental; assessment
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Language

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy individuals: No intervention
  Healthy participants ages 14-32 for a neuroimaging study.
- Individuals with Autism Spectrum Disorder: No intervention
  ASD participants ages 14-32 for a neuroimaging study.

SUMMARY:
The purpose of this study is to create a subject database to recruit for current and future studies in research on autism and other neurodevelopmental disabilities.

DETAILED DESCRIPTION:
Aim 1: to recruit people interested in research on autism and other neurodevelopmental disabilities

Aim 2: to complete a diagnostic assessment, to confirm the diagnosis of autism spectrum disorder or other developmental disability (e.g., developmental language delay) in our patient population and rule out a diagnosis of autism spectrum disorder and other comorbid conditions in our control group

Aim 3: to maintain subject information in a database, from which we can recruit for our studies

ELIGIBILITY:
Inclusion Criteria:

* Typically-developing, healthy adolescents and adults (ages 14-32)
* Adolescents and adults with autism spectrum disorder (ages 14-32)

Exclusion Criteria:

* Extreme premature birth (<34 weeks)
* Known genetic disorders related to autism (e.g. Fragile X)
* Recent diagnosis of psychosis (within 6 months)
* Some other psychiatric diagnoses may be excluded following screening (e.g. Tourette's syndrome).
* Metal implants / permanent retainers / hair dyes with metallic components

Ages: 14 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adult/Pediatric
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Kenet, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Martinos Center of Biomedical Imaging, Charlestown, Massachusetts, United States